CLINICAL TRIAL: NCT01911377
Title: The Efficacy of Botulinum Toxin Type A in the Treatment of Allodynic-Type Neuropathic Pain in People With Spinal Cord Injury or Multiple Sclerosis
Brief Title: Botulinum Toxin Type A for Treating Allodynic Pain in SCI and MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 12 SCI volunteers completed the study. As the data analysis was negative, the decision was made not to proceed with MS recruitment.
Sponsor: University of Manitoba (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Director, Spinal Cord Injury Rehabilitation Program, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Botox 2013
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Neuropathic Pain; Allodynia
MeSH Terms: conditions — Neuralgia; Hyperalgesia | interventions — Botulinum Toxins, Type A; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Botulinum Toxin Type A (Active Comparator): 200 units of Botulinum Toxin Type a will be administered intradermally to the allodynic area chosen for study.The allodynic area will be mapped, and the number of injections needed to cover the allodynic area without exceeding 40 injection sites will be determined.
  All participants will receive a cream formulation of lidocaine and prilocaine (EMLA) applied to the painful area 60 minutes before the injections to minimize any discomfort caused by the injections.
  Interventions: Drug: Botulinum Toxin Type A
- Arm 2: Normal Saline for Injection (Placebo Comparator): Normal saline for intradermal injection will be prepared by the Investigational Pharmacy in a manner as to be indistinguishable from active drug. The allodynic area will be mapped so as to determine the number of injections needed to cover the whole allodynic area without exceeding 40 injection sites. All participants will receive a cream formulation of lidocaine and prilocaine (EMLA) applied to the painful area 60 minutes before the injections to minimize any pain caused by the injections.
  Interventions: Drug: Normal Saline for Injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Arms: Arm 1: Botulinum Toxin Type A
Drug: Normal Saline for Injection
  Arms: Arm 2: Normal Saline for Injection

SUMMARY:
This study will examine the efficacy of Botulinum Toxin Type A ("Botox") in treating Allodynic-type neuropathic pain in people with spinal cord injury or multiple sclerosis.

Neuropathic pain is pain initiated or caused by injury to or disease of the nervous system, and is common in spinal cord injury patients or people with multiple sclerosis.

Allodynia is a type of neuropathic pain caused by something that normally would not cause pain, such as light touch, pressure from clothing, or bed sheets brushing against the skin.

Botox has been used to treat the muscle overactivity that causes spasticity in spinal cord injured patients. It has been noticed to exert some analgesic(pain relieving) effect, and has recently been studied as a treatment for neuropathic pain.

We want to see if Botox, injected intradermally, will relieve the symptoms of allodynic-type neuropathic pain.

24 volunteers are to be enrolled, with 16 receiving active treatment, and 8 "controls" receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the criteria for neuropathic pain causing allodynia according to IASP pain terminology.
* Allodynia that is resistant to, or has failed, the standard level of care measures for more that six months.
* Allodynia pain on a daily basis.
* Allodynia pain that scores at least 4/10 on a pain numerical scale.
* Other pain medications(including antidepressants and anticonvulsants)have been maintained at a stable dose for at least 2 months prior to enrollment.
* Ability to communicate in English.

Exclusion Criteria:

* Presence of other pain syndromes (e.g.,fibromyalgia, ongoing peripheral neuropathic pain.
* Allergy to Botulinum Toxin Type A.
* Allergy to albumin.
* Use of Botulinum Toxin Type A for other treatment indications in the 3 months prior to enrollment.
* Renal failure.
* Hepatic failure.
* Neuromuscular junction disorders.
* Bleeding diathesis.
* Cognitive impairment, dementia, major depression or psychotic disorder.
* Pregnant or breastfeeding.
* Infection at the injection site.
* Active alchohol or substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Baseline and daily until study completion at 13 weeks
  The primary outcome measure will be the self-reported average pain intensity from each morning's record in a diary. The average(self-reported) pain intensity will be measured at the screening visit, then the daily diary will be dispensed. The diary will ask for the average pain intensity of the last 24 hours using an 11-point numerical scale, with 0 representing no pain and 10 representing the worst pain imaginable

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | Baseline and follow-up visits(at weeks 1, 4, 8 and 13)
  This scale rates the mean intensity of 10 neuropathic pain symptoms and their combination into 5 distinct dimensions during the last 24 hours on an 11-point (0-10) numerical scale
The Hospital Anxiety and Depression Scale | Baseline and follow-up visits (at weeks 1, 4, 8 and 13).
  14 items scored as anxiety and depression
Daily Sleep Interference Scale | Baseline and daily during study period until week 13.
  Asks if pain interfered with sleep in the past 24 hours,using an 11-point scale (O-pain did not interfere with sleep, 10-pain completely interfered with sleep).
  Dispensed at baseline.
Clinician Global Impression Scale | Final visit at week 13
  Assesses the clinician's impression of Efficacy and Tolerability of study medication using a 4-point scale, with 1 being Very good, and 4 being Poor
Patient's Global Impression Scale | Final visit at week 13
  Measures the patients global impression of the efficacy and tolerability of the study medication on a 4-point scale, with 1 representing very good, and 4 representing poor

OTHER OUTCOMES:
Measurement of brush-induced allodynia | Baseline and follow-up visits(weeks 1, 4, 8 and 13)
  The area of skin with allodynic pain is stroked with a standardized brush and the patient reports any pain associated with the stroking.
Measurement of mechanical sensations and pain thresholds | Baseline and follow-up visits (weeks 1, 4 , 8 and 13)
  An algometer (a device that pushes against the skin to measure when pain is felt) will be used on the allodynic area
Recording Area of allodynia | Baseline and follow-up visits (at weeks 1, 4, 8 and 13)
  The area of allodynic pain to be treated is traced on transparent paper
Measurement of temperature sensations and pain thresholds | Baseline and follow-up visits(at weeks 1, 4, 8 and 13)
  A thermo-test is used to measure temperature sensations and pain thresholds in the allodynic area

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ethans, MD, Principal Investigator — Health Sciences Centre
Locations (1):
- WRHA Health Sciences Centre Rehabilitation Hospital, Winnipeg, Manitoba, Canada